CLINICAL TRIAL: NCT01319214
Title: Reconsolidation as a Treatment Target for Cocaine Addiction
Brief Title: Reducing Drug Craving Memories
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Marco Leyton, MUHC
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 10-039-PSY
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-01

CONDITIONS: Cocaine Addiction
Keywords: cocaine addiction treatment craving
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Inderal, neutral cues (Experimental)
  Interventions: Drug: Inderal
- Inderal, drug cues (Experimental)
  Interventions: Drug: Inderal
- Placebo, neutral cues (Experimental)
  Interventions: Drug: Inderal
- Placebo, drug cues (Experimental)
  Interventions: Drug: Inderal

INTERVENTIONS:
Drug: Inderal — Inderal vs. placebo will be administered with or without cocaine cues

SUMMARY:
The primary objective is to investigate the potential ability of Inderal (propranolol hydrochloride) to diminish the reconsolidation of motivationally potent drug-related cues in cocaine dependent participants. If effective in this laboratory model, Inderal may have clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 60 psychotropic medication-free men or women (15 subjects x 4 groups) who have met DSM-IV-TR diagnostic criteria for cocaine dependence for the past 6 months (age 18 - 50 years old);
* Minimum of three days cocaine abstinent on study days;
* Primary use of cocaine is intra-nasal or smoked crack

Exclusion Criteria:

* Medical conditions that might be aggravated by participation in the study:

  * cardiovascular disorders that might be aggravated by participation in the study: hypotension (SBP: < 100 mmHg), bradycardia (heart rate < 60 /min), severe atrioventricular block (Type II or III), severe hypertension (SBP: > 160 mmHg; DBP: > 100 mmHg), myocardial infarction, history of chest pain and admission to ED for chest pain;
  * respiratory disorders: bronchial asthma and chronic obstructive pulmonary disease;
  * diabetic patients treated with insulin or oral hypoglycemic agents. Propranolol may mask the first signs of a developing hypoglycemia.
* Seropositive pregnancy test
* Comorbidity with current axis I psychiatric disorders other than anxiety, affective and substance use disorders
* Severe liver disfunction
* Current or recent (< 5 half lives) use of medications that may interact with Inderal (see above)
* Positive urine tox screen for barbiturates. Positive breath alcohol screen. {Note: all urine tox screen results will be destroyed immediately after collection. The information will not be stored}

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Self-report drug craving | One day and one month post-treatment
  One day and one month after the intervention, the investigators will measure drug craving using visual analog scales (VAS) and the Cocaine Craving Questionnaire (CCQ).

SECONDARY OUTCOMES:
Drug use | One month after the intervention
  One month after the intervention, participants will be interviewed about their drug and alcohol use